CLINICAL TRIAL: NCT05528237
Title: Advancing Cervical Cancer Screening Through Self-Sampling (ACCESS): A Pilot Study of HPV Self-sampling for Cervical Cancer Prevention in Washington State
Brief Title: HPV Self-sampling to Improve Access to Cervical Cancer Screening for Persons With HIV and/or Underserved Individuals
Acronym: ACCESS
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: Principal Investigator, Darcy W Rao, PhD, Acting Assistant Professor: School of Public Health, University of Washington
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: STUDY00014442; 5KL2TR002317-05 (NIH)
Record Dates: First submitted 2022-08-29; First posted 2022-09-06 (Actual); Last update posted 2022-09-06 (Actual); Status verified 2022-08

CONDITIONS: Cervical Cancer
Keywords: Screening; Self-collection; Self-sampling; Cervical cancer; HPV; HIV
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- HPV self-sampling (Experimental): Participants will be offered self-collection kits for HPV-based cervical cancer screening.
  Interventions: Device: Flocked swab paired with Roche Cobas 4800

INTERVENTIONS:
Device: Flocked swab paired with Roche Cobas 4800 — Consenting individuals will insert the sterile flocked swab into the vagina, rotate at least once, and store in the provided dry tube. The sample will be stored at ambient temperature and routed to the lab for HPV testing with Roche Cobas 4800.
  Other Names: COPAN 552c FLOQSwabs

SUMMARY:
The objective of this study is to evaluate self-collection of vaginal samples for HPV testing as an alternative cervical cancer screening strategy for persons with HIV and/or limited access to care. Self-collection kits will be offered to persons who refuse a Pap smear or are overdue (>=6 months) for cervical cancer screening, with screening uptake recorded as a primary outcome. Kits will be offered in-clinic to individuals who refuse a Pap smear, and individuals overdue for screening will have the option to receive and return kits in the mail. The investigators will additionally administer a phone-based survey to evaluate knowledge about HPV and cervical cancer, barriers and facilitators to screening, and attitudes towards screening. Data from medical records will be abstracted to describe the clinical characteristics of the sample and measure receipt of follow-up procedures. Focus groups will be conducted with clinic administrators, staff, and HIV and women's health experts to evaluate clinic and provider barriers and facilitators to cervical cancer screening. The investigators hypothesize that HPV self-sampling will result in favorable patient-centered outcomes and could reduce disparities in access to screening.

ELIGIBILITY:
Inclusion Criteria:

* Age >=25 and <65 (individuals without diagnosed HIV) or >=30 years (individuals with diagnosed HIV)
* Female sex at birth
* Proficient in English or Spanish
* Refused a Pap smear or are >=6 months overdue for cervical cancer screening

Exclusion Criteria:

* Current pregnancy
* Complete hysterectomy
* History of cervical cancer
* Unable to provide informed consent

Min Age: 25 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-08-18 (Actual); Primary Completion 2022-09-30 (Estimated); Study Completion 2022-10-07 (Estimated)

PRIMARY OUTCOMES:
Proportion of eligible individuals who accept self-sampling kits | Baseline (during clinical and/or study recruitment encounter)
  the proportion of eligible individuals due or overdue for screening who agree to collect a vaginal sample for HPV testing.
Proportion of eligible individuals who submit self-sampled specimens | 3 weeks from enrollment
  the proportion of individuals who agree to self-collection who return samples
Satisfaction with self-collection | Within 2 weeks of sample collection
  Participants will use a 5-point Likert scale (strongly agree, agree, neutral, disagree, strongly disagree) to respond to the statement, "I was satisfied with the self-collection experience."
Confidence with self-collection | Within 2 weeks of sample collection
  Participants will use a 5-point Likert scale (strongly agree, agree, neutral, disagree, strongly disagree) to respond to the statement, "I am sure I got a good sample using the swab."
Recommendation of self-collection | Within 2 weeks of sample collection
  Participants will use a 5-point Likert scale (strongly agree, agree, neutral, disagree, strongly disagree) to respond to the statement, "I would recommend self-collection to a friend."
Ease of returning home kits | Within 2 weeks of sample collection
  Participants who collected a sample at home will use a 5-point Likert scale (strongly agree, agree, neutral, disagree, strongly disagree) to respond to the statement, "It was easy to return my sample (by mail or to the clinic)."

SECONDARY OUTCOMES:
Proportion of eligible individuals who return samples with adequate specimens | 3 weeks from enrollment
  the proportion of returned samples that have valid specimens for HPV testing
Knowledge about HPV and cervical cancer screening | Baseline
  a survey to measure participant's knowledge about HPV and cervical cancer screening
Perceived risk of cervical cancer | Baseline
  a survey to measure participant's perceived risk of cervical cancer
Attitudes and preferences for screening | Baseline
  a survey to measure participant's attitudes and preferences for cervical cancer screening
HPV prevalence checklist | Baseline
  the distribution of HPV results from all individuals who return a self-sampled specimen
Receipt of follow-up care | Up to 6 months after self-sampling
  Among participants who screen positive for hrHPV, measure the proportion who receive indicated follow-up care (cytology and/or colposcopy)
Reflex cytology results checklist | Up to 6 months after self-sampling
  the results of cytology tests following positive self-sampled HPV results
Colposcopy results checklist | Up to 6 months after self-sampling
  the results of colposcopy tests following positive self-sampled HPV results.
Provider and/or clinic barriers and facilitators to cervical cancer screening survey | During study year 1
  focus group discussions with clinic administrators, staff and other HIV and women's health experts. These discussions will cover: barriers to clinician-administered screening (i.e., Pap screening and clinician-collected HPV samples); perceived patient barriers to clinician-administered screening and follow-up procedures; perceived facilitators to cervical cancer screening and follow-up; and feasibility of offering HPV self-sampling kits as a potential primary screening strategy.

CONTACTS AND LOCATIONS:
Overall Officials: Darcy Rao, PhD, MPH, Principal Investigator — University of Washington
Locations (3):
- United States (3):
  - SHE Clinic, Seattle, Washington
  - Madison Clinic, Seattle, Washington
  - MAX Clinic, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Yes
De-identified study data will be posted on a repository for use in studies on access to healthcare and sexual and reproductive health, including but not limited to cervical cancer services.
Time Frame: Data will be available within 6 months of study end date.
Access Criteria: Investigators interested in using study data will need to contact the investigator and sign a data use agreement.